CLINICAL TRIAL: NCT06541639
Title: A Dose Escalation and Expansion Study to Evaluate the Safety, Tolerability, Immunogenicity, and Initial Efficacy of EVM16 Injection As a Single and Combination with Tislelizumab in Subjects with Advanced or Recurrent Solid Tumors
Brief Title: EVM16 Injection As a Single and Combination with Tislelizumab in Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Peking University (Other)
Collaborators: Shanghai Cancer Centre (Other); Everest Medicines (China) Co.,Ltd. (Industry)
Responsible Party: Principal Investigator, Shen Lin, Beijing Cancer Hospital, Peking University Cancer Hospital & Institute
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: EVM16CX01
Record Dates: First submitted 2024-07-29; First posted 2024-08-07 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Advanced or Recurrent Solid Tumors
Keywords: solid tumor; tumor vaccine; immune checkpoint inhibitor
MeSH Terms: interventions — tislelizumab

STUDY DESIGN:
Intervention Model Description: A Dose Escalation and Expansion Study to Evaluate the Safety, Tolerability, Immunogenicity, and Initial Efficacy of EVM16 Injection as a Single and Combination with Tislelizumab in Subjects with Advanced or Recurrent Solid Tumors.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Dose Escalation Level 1 (Experimental): EVM16 dose level 1 as single and combined therapy with Tislelizumab.
  Interventions: Biological: EVM16; Drug: Tislelizumab
- Dose Escalation Level 2 (Experimental): EVM16 dose level 2 as single and combined therapy with Tislelizumab.
  Interventions: Biological: EVM16; Drug: Tislelizumab
- Dose Escalation Level 3 (Experimental): EVM16 dose level 3 as single and combined therapy with Tislelizumab.
  Interventions: Biological: EVM16; Drug: Tislelizumab
- Dose Expansion (Experimental): EVM16 RP2D dose in combination with Tislelizumab.
  Interventions: Biological: EVM16; Drug: Tislelizumab

INTERVENTIONS:
Biological: EVM16 — cancer vaccine
Drug: Tislelizumab — Anti-PD1 antibody
  Other Names: Tevimbra

SUMMARY:
The goal of this clinical trial is to learn the side effects, safety and effect of a tumor vaccine (EVM16) alone or in combined with an anti-PD-1 antibody (tislelizumab) . This clinical trial will include solid tumor patients who failed standard treatment.

The main questions to answer are:

Safety of EVM16. Suitable dose of EVM16. Effects of EVM16 combined with tislelizumab.

ELIGIBILITY:
Key Inclusion Criteria:

* Recurrent or metastatic solid tumors that have been histologically or cytologically pathologically confirmed and are not amenable to radical treatment with surgery or local therapy.
* Patients with advanced or recurrent solid tumors who have failed prior standard therapy.
* Expected survival period >6 weeks at the time of informed consent.
* Adequate organ function
* Eastern Cooperative Oncology Group (ECOG) Physical Status Score 0 to 1.
* Is willing to provide archival or fresh tumor tissue samples for EVM16 production.
* Has adequate treatment washout period prior to first study dose.
* Has at least one measurable lesion as assessed by the investigator according to RECIST version 1.1 criteria before enrollment.

Key Exclusion Criteria:

* Primary central nervous system (CNS) malignancies that are symptomatic, untreated, or in need of curative treatment, or subjects with CNS metastases.
* Uncontrolled co-morbidities.
* Cerebrovascular event (stroke, transient ischemic attack, etc.) within 4 months prior to the signing of inform consent form.
* In screening period male QTcF interval >450 ms; Female QTcF interval >470 ms (calculated by the Fridericia formula).
* Left ventricular ejection fraction (LVEF) < 50% during the screening period.
* Diagnosis of immunodeficiency, or history or syndrome of active as well as former autoimmune disease with risk of relapse, or a disease requiring systemic steroid hormone or immunosuppressive drug therapy.
* Subjects with a history of positive human immunodeficiency virus (HIV) test or acquired immunodeficiency syndrome (AIDS).
* Co-infection HBV and HCV.
* Presence of any active infection requiring systemic therapy.
* Patients who are still on any other investigational medications treatment at the time of screening.
* Previous treatment with cell therapy, tumor vaccines, cytokines, or growth factors for cancer control.
* Patients with prior intolerance to tislelizumab resulting in permanent termination of tislelizumab.
* History or presence of significant lung disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2025-03-04 (Actual); Primary Completion 2028-03-31 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
safety and tolerability | From the first study intervention to 90 days after the last study intervention.
  The incidence and severity of adverse events (AEs) and serious adverse events (SAEs), the incidence of dose-limiting toxicity (DLT) （only in phase Ia）, and the incidence of AEs of grade 3 or higher were assessed according to the NCI CTCAE v5.0 in the treatment of EVM16 alone as well as EVM16 in combination with Tislelizumab.
RP2D for EVM16 | During the intervention, up to approximately 1 year.
  Based on safety, tolerability, immunogenicity to determine RP2D.

SECONDARY OUTCOMES:
immunogenicity of EVM16 | during the intervention, up to 1 year
  Based on proportion of IFN-γ-positive T cells and/or T cell receptor sequences after EVM16 administration to assess the immunogenicity of EVM16 in subjects with advanced or recurrent solid tumours.
objective response rate (ORR) of EVM16 in combination with tislelizumab | From date of first study dose until the date of disease progression, or until the patient start subsequent anti-cancer treatment, or death, or lost to follow up or the study ends, whichever occurs first.
  Proportion of patients with partial response (PR) and complete response (CR) as assessed by the investigators according to RECIST v1.1 in EVM16 combined with tislelizumab arm.
disease control rate (DCR) of EVM16 in combination with tislelizumab | From date of first study dose until the date of disease progression, or until the patient start subsequent anti-cancer treatment, or death, or lost to follow up or the study ends, whichever occurs first.
  Proportion of patients with partial response (PR) , complete response (CR) and stable disease (SD) as assessed by the investigators according to RECIST v1.1 in EVM16 combined with tislelizumab arm.
duration of disease remission (DOR) of EVM16 in combination with tislelizumab | From date of first study dose until the date of disease progression, or until the patient start subsequent anti-cancer treatment, or death, or lost to follow up or the study ends, whichever occurs first.
  Duration of objective response (PR and CR) as assessed by the investigators according to RECIST v1.1 in EVM16 combined with tislelizumab arm.
time to remission (TTR) of EVM16 in combination with tislelizumab | From date of first study dose until the date of disease progression, or until the patient start subsequent anti-cancer treatment, or death, or lost to follow up or the study ends, whichever occurs first.
  Time from enrollment to objective response (PR and CR) as assessed by the investigators according to RECIST v1.1 in EVM16 combined with tislelizumab arm.
PFS of EVM16 in combination with tislelizumab （Only in phase Ib） | From date of first study dose until the date of disease progression, or until the patient start subsequent anti-cancer treatment, or death, or lost to follow up or the study ends, whichever occurs first
  Progression-free survival (PFS) as assessed by the investigators according to RECIST v1.1 in EVM16 combined with tislelizumab arm.

CONTACTS AND LOCATIONS:
Overall Officials: Lin Shen, MD, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (2):
- China (2):
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No